CLINICAL TRIAL: NCT04338230
Title: The Effect of Progressive Muscle Relaxation on Depression and Adaptation to Old Age of Elderly Women: A Randomized Controlled Trial
Brief Title: Progressive Muscle Relaxation and Adaptation to Old Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University (Other)
Responsible Party: Principal Investigator, İlknur Gökşin, PhD, Assistant Professor, Aksaray University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/245
Record Dates: First submitted 2020-04-04; First posted 2020-04-08 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Elderly Women
Keywords: Relaxation exercises; Elderly; Women; Adaptation to old age

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Experimental group (Experimental): Women aged 65 and over (the standardized Mini-Mental State Examination (MMSE) test cognitive levels score of 23 and above points). Progressive muscle relaxation exercises are applied to the intervention group as 30-minute sessions three times a week for eight weeks.
  Interventions: Other: Progressive muscle relaxation exercise
- No Intervention: Control group (No Intervention): Women aged 65 and over (the standardized Mini-Mental State Examination (MMSE) test cognitive levels score of 23 and above points).

INTERVENTIONS:
Other: Progressive muscle relaxation exercise — "Relaxation Exercises CD Audio Records" prepared by Turkish Psychological Association is used. Before starting the PMR exercises, the woman in the intervention group is provided to lie on a comfortable seat or bed, stretching the muscles of the face and all body for about 10 seconds starting from the hands to the foot in line with the sound recordings of the PKG exercises and then holding the deep breath while each muscle group is stretching, It is applied as a slow release of this breath during relaxation. In this way, the muscle groups in the hands, arms, neck, shoulders, chest, abdomen, hips, feet and fingers, the face and the whole body are tensioned and relaxed, and the woman is relaxed. During the eight-week period, the women are called by the researcher once a week and the exercises are reminded. Home visit There are 2 home visits at week 1 and at week 8. In case of need, repeated home visits are provided to ensure the continuity of the application.
  Arms: Experimental: Experimental group

SUMMARY:
Changes and limitations in the aging process affect adaptation to old age. It is important for women to adapt to the problems of old age, find a solution and cope. This study was aimed to determine the effect of progressive muscle relaxation exercises on the level of depression and adaptation to old women.

DETAILED DESCRIPTION:
The aging process is considered as a result of the decline observed in basic cognitive functions such as attention, perception, memory, and causes problems in the communication of the elderly with the environment. For these problems, it affects the adaptation of the elderly in his environment and himself.

There are a limited number of studies in the literature to increase the adaptation of older individuals to old age. In the studies in the literature, it was stated that the rate of depression is higher in female individuals, and being male and having a high education level positively affect the adaptation of individuals to old age. In a national study, it was determined that as age increases, adaptation to old age decreases.

Progressive muscle relaxation (PMR), one of the nonpharmacological methods, involves the voluntary stretching and relaxation of large muscle groups (hand-starting, foot-end muscle groups) in the human body. It is known that PMR exercises are frequently used in nursing research because of the effects of reducing anxiety and fatigue and improving sleep quality, and reducing nausea-vomiting. However, no study was found on the effect of depression and adaptation to old age. Due to these positive effects of PMR determined in the literature, it is thought that elderly women can positively affect their levels of depression and adaptation to old age.

Objective: Evaluate the effects of progressive muscle relaxation on the depression and adaptation of elderly women to aging.

Methodology: This is randomized clinical test. The sample was made up of 49 elderly women who applying to the family health center (21 in the experimental group and 28 in control group). The progressive muscle relaxation was employed. In order to collect the data, we adopted the interview with form filling technique, using the introductory information form, Assessment Scale of Adaptation Difficulty for the Elderly (ASADE) and Geriatric Depression Scale Short Form (GDS-S). Progressive muscle relaxation will be performed for a total of 8 weeks, 3 days a week, for 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and above,
* Do not have a diagnosis of dementia and psychiatric disease by the doctor and have a mini-mental test score of 23 and above,
* Being independent in practicing daily living activities
* There is no problem with communication

Exclusion Criteria:

* Under the age of 65
* Being addicted in daily life activities
* Being diagnosed with dementia and psychiatric illness
* Mini-mental test score below 23

Ages: 65 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Standardized Mini Mental Test (SMMT) | Pretest of study
  SMMT evaluates cognitive status. Women with a SMMT score 23 and above (min.0 - max. 30) were included in the study.

SECONDARY OUTCOMES:
Geriatric Depression Scale-Short Form (GDS-SF) | 2 month
  Evaluation of depressive symptoms of elderly individuals. In the evaluation of the scale, the answers to no, positive questions and yes to negative questions were matched by 1 point. A total score of 6 and above is considered significant for the diagnosis of depression.
Assessment Scale of Adaptation Difficulty for the Elderly | 2 month
  The difficulties in adaptation to old age of elderly individuals were evaluated using the Assessment Scale of Adaptation Difficulty for the Elderly (ASADE). The scores obtained from the items of the scale (24 ıtems) are collected and divided by the number of questions to obtain the total score of the scale. The level of adaptation to old age decreases as the score obtained from the scale by an individual increases. ASADE total score min. 0- max. 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Aksaray University, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No